CLINICAL TRIAL: NCT04770870
Title: Post Approval Study 2: Hintermann Series H3 Total Ankle Replacement System
Brief Title: Post Approval Study2: Hintermann Series H3 Total Ankle Replacement System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DT MedTech, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAS 002
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis Ankle; Post-Traumatic Osteoarthritis of Ankle; Osteoarthritis of Ankle Secondary to Inflammatory Arthritis (Disorder)

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single arm post approval study of 232 subjects up to 10 US study sites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Other): All subjects who meet eligibility, consented, and enrolled into the study will receive treatment.
  Interventions: Device: Hintermann Series H3 Total Ankle Replacement System

INTERVENTIONS:
Device: Hintermann Series H3 Total Ankle Replacement System — Intervention will include receiving the FDA approved Hintermann Series H3 Total Ankle Replacement System, to include a tibial component, a polyethylene inlay, and a talar component.

SUMMARY:
The H3 TAR Prosthesis was approved by FDA (P160036) on June 4, 2019. Continued approval of the premarket approval application (PMA) is contingent upon the submission of periodic reports (Annual Report), required under 21 CFR 814.84. In order to provide continued reasonable assurance of the safety and effectiveness of the PMA device, data from this post-approval study must be submitted to FDA in a PMA Post-Approval Study Report per the requirements set forth in the approval.

DETAILED DESCRIPTION:
The Hintermann Series H3® (H3) prosthesis is a mobile bearing total ankle replacement (TAR) indicated for use as a non-cemented implant to replace a painful arthritic ankle joint due to primary osteoarthritis, post-traumatic osteoarthritis or arthritis secondary to inflammatory disease (e.g., rheumatoid arthritis, hemochromatosis, etc.).

The present version (third generation) of the H3 TAR and the earlier generations of this total ankle system have been marketed (initially in 2003) under a license agreement in Europe, South Korea, Australia, and Canada and other countries outside the U.S. (OUS). The H3 TAR prosthesis has been used in over 20,000 procedures in the markets OUS. The H3 TAR device has not been withdrawn from marketing for any reason.

The H3 TAR Prosthesis was approved by FDA (P160036) on June 4, 2019. Continued approval of the premarket approval application (PMA) is contingent upon the submission of periodic reports (Annual Report), required under 21 CFR 814.84. In order to provide continued reasonable assurance of the safety and effectiveness of the PMA device, data from this post-approval study must be submitted to FDA in a PMA Post-Approval Study Report per the requirements set forth in the approval.

ELIGIBILITY:
Inclusion Criteria:

* Each potential subject must be an appropriate candidate for mobile bearing TAR by having: a primary osteoarthritis, post-traumatic osteoarthritis, or arthritis secondary to inflammatory disease, as determined by the Principle Investigator.
* Willingness to participate in the study and follow-up visits
* Written informed consent, including authorization to release collected health data

Exclusion Criteria:

* Skeletal immaturity
* Bone stock inadequate to support the device including:

  * Severe osteoporotic or osteopenic condition or other conditions resulting in poor bone quality
  * Avascular necrosis of the talus
* Active or prior deep infection in the ankle joint or adjacent bones
* Malalignment or severe deformity of involved or adjacent anatomic structures including:

  * Hindfoot or forefoot malalignment precluding plantigrade foot
  * Significant malalignment of the knee joint
  * Insufficient ligament support that cannot be repaired with soft tissue stabilization (syndesmosis disruption)
* Charcot joint or peripheral neuropathy that may lead to Charcot joint of the affected ankle
* Neuromuscular disease resulting in lack of normal muscle function about the affected ankle
* Lower extremity vascular insufficiency demonstrated by Doppler arterial pressure
* Poor skin and soft tissue quality about the surgical site
* Immunosupressive therapy
* Prior ankle fusion or revision of total ankle replacement
* High demanding sport activities (e.g., contact sports, jumping)
* Suspected or documented metal allergy or intolerance
* Condition or situation which, in the Physician's opinion, puts the subject at significant risk, or may interfere significantly with the subject's participation in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Measurement | 5-years
  The Primary Safety Measurement for this study is the percentage of patient subjects with a serious device-related adverse event, other than a revision or removal within 2 years.
Primary Effectiveness Measurement | 5-years
  The co-primary effectiveness measurements for this study are the American Orthopaedic Foot and Ankle Society (AOFAS) score at 2 years or more, the survivorship (absence of removal/revisions of metal components) within 5 years post-surgery, and the percentage of subjects with a serious device-related adverse event, other than a revision or removal within 2 years.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Los Angeles Institute of Foot and Ankle Surgery, Mission Hills, California
  - Florida Orthopedic Foot & Ankle Center, Sarasota, Florida
  - Paley Orthopedic & Spine Institute, West Palm Beach, Florida
  - Orthopaedic Associates, Evansville, Indiana
  - Department of Orthopedic Surgery, Johns Hopkins Outpatient Center, Baltimore, Maryland
  - New Mexico Bone and Joint Institute, Alamogordo, New Mexico
  - Duke Orhtopaedics Arringdon, Morrisville, North Carolina
  - Dept. of Orthopedic Surgery and Rehabilitation, University of Oklahoma, Oklahoma City, Oklahoma
  - MUSC Department of Orthopaedics/Foot and Anke Services, Charleston, South Carolina
  - Spring Branch Podiatry, PLLC, Houston, Texas

IPD SHARING:
Plan to Share IPD: No